CLINICAL TRIAL: NCT01170494
Title: Effect of Vitamin D Oral Supplements on 25 OH Vitamin D Levels: A Randomized Controlled Trial
Brief Title: Effect of Vitamin D Oral Supplements on 25 OH Vitamin D Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Muhammad Maher Hammami, Chairman, Department of Clinical Studies & Empirical Ethics, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAC 2101041
Record Dates: First submitted 2010-07-25; First posted 2010-07-27 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D2, vitamin D3, 25 Oh vitamin D2, 25 Oh vitamin D3
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- D2 2000 IU daily (Active Comparator)
  Interventions: Drug: ergocalciferol 2000 IU orally, daily
- D3 2000 IU daily (Active Comparator)
  Interventions: Drug: cholecalciferol 2000 IU orally daily
- D2 1000 IU + D3 1000 IU daily (Active Comparator)
  Interventions: Drug: ergocal1000 IU & cholecal 1000 IU orally daily
- D2 25000 IU Q2wk (Active Comparator)
  Interventions: Drug: ergocalciferol 25000 IU oraly every 2 weeks
- D3 25000 IU Q2wk (Active Comparator)
  Interventions: Drug: Cholecalciferol 25000 IU orally every 2 weeks
- D2 50000 IU Q4wk (Active Comparator)
  Interventions: Drug: ergocalciferol 50000 IU orally every 4 weeks
- D3 50000 IU Q4wk (Active Comparator)
  Interventions: Drug: Cholecalciferol 50000 orally every 4 weeks
- placebo daily (Placebo Comparator)
  Interventions: Drug: placebo orally everyday

INTERVENTIONS:
Drug: ergocalciferol 2000 IU orally, daily — ergocalciferol 2000 IU orally, daily
  Other Names: ergocalciferol
  Arms: D2 2000 IU daily
Drug: ergocalciferol 25000 IU oraly every 2 weeks — ergocalciferol 25000 IU oraly every 2 weeks
  Other Names: ergocalciferol
  Arms: D2 25000 IU Q2wk
Drug: ergocalciferol 50000 IU orally every 4 weeks — ergocalciferol 50000 IU orally every 4 weeks
  Other Names: ergocalciferol
  Arms: D2 50000 IU Q4wk
Drug: ergocal1000 IU & cholecal 1000 IU orally daily — ergocalciferol 1000 IU and cholecalciferol 1000 IU orally every day
  Other Names: ergocalciferol and cholecalciferol
  Arms: D2 1000 IU + D3 1000 IU daily
Drug: cholecalciferol 2000 IU orally daily — cholecalciferol 2000 IU orally everyday
  Other Names: cholecalciferol
  Arms: D3 2000 IU daily
Drug: Cholecalciferol 25000 IU orally every 2 weeks — Cholecalciferol 25000 IU orally every 2 weeks
  Other Names: Cholecalciferol
  Arms: D3 25000 IU Q2wk
Drug: Cholecalciferol 50000 orally every 4 weeks — Cholecalciferol 50000 orally every 4 weeks
  Other Names: Cholecalciferol
  Arms: D3 50000 IU Q4wk
Drug: placebo orally everyday — placebo orally everyday
  Other Names: placebo
  Arms: placebo daily

SUMMARY:
Vitamin D deficiency is common world wide. 25 OH vitamin D level is the best indicator of vitamin D status. Vitamin D supplements are available as vitamin D2 or D3, in small daily or large weekly/monthly doses. Controversy continues on the relative potency of vitamin D2 compared to D3 and of daily compared to weekly or monthly doses, in increasing/maintaining total 25 OH vitamin D level.

The investigators plan to conduct a controlled trial to compare the effect of various vitamin D supplements on 25 OH vitamin D levels in healthy adults with starting 25 OH vitamin D level between 20 to 50 nmol/L.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults living in Riyadh area who consume no more than one serving of milk/day, do not take vitamin supplement, habitually have less than 10 hr of sun exposure per week, don't suffer from granulomatous conditions, liver disease, or kidney disease, and don't take anticonvulsants, barbiturates, or steroids.
* 25 OH vitamin D level between 20 to 50 nmol/L.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
area under the curve of 25 OH vitamin D level | 140 days
  area under the curve of total 25 OH vitamin D level from day 1 to 140

SECONDARY OUTCOMES:
Cmax of 25 OH vitamin D | 140 days
  Cmax of total 25 OH vitamin D over the treatment period of 140 days
Tmax of 25 OH vitamin D level | 140 days
  Tmax of total 25 OH vitamin D over the treatment period of 140 days
area under the curve of vitamin D level | 140 days
  area under the curve of total vitamin D level over 140 days
incidence of hypercalcemia | 140 days
incidence of hypercalciuria | 140 days

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad M Hammami, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- King Faisal Specialist Hospital & research Center, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Hammami MM, Yusuf A. Differential effects of vitamin D2 and D3 supplements on 25-hydroxyvitamin D level are dose, sex, and time dependent: a randomized controlled trial. BMC Endocr Disord. 2017 Feb 24;17(1):12. doi: 10.1186/s12902-017-0163-9. PMID 28231782